CLINICAL TRIAL: NCT01931371
Title: An Outcome and Cost Analysis of Anal Fistula Plug Versus Endorectal Advancement Flap in Complex Anal Fistulae
Brief Title: Anal Fistula Plug Versus Endorectal Advancement Flap
Acronym: AFPERAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFPERAF; KEK-ZH-Nr. 2013-XYZ (Other: Cantonal Ethical Committee Canton of Zurich)
Record Dates: First submitted 2013-08-05; First posted 2013-08-29 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Anal Fistula
Keywords: fistula in ano; anal fistula; recurrence; costs
MeSH Terms: conditions — Rectal Fistula; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recurrent anal fistula (Active Comparator): Patients with a complex anal fistula that recurred after surgery with an Anal Fistula Plug or and Endorectal Advancement Flap
  Interventions: Procedure: Anal Fistula Plug; Procedure: Endorectal Advancement Flap
- No recurrence of anal fistula (Active Comparator): Patients with a complex anal fistula that did not develop recurrence after surgery with an Anal Fistula Plug or and Endorectal Advancement Flap
  Interventions: Procedure: Anal Fistula Plug; Procedure: Endorectal Advancement Flap

INTERVENTIONS:
Procedure: Anal Fistula Plug — Surgical procedure for the treatment of anal fistula with an Anal Fistula Plug
  Other Names: Anal Fistula Plug (Cook Medical Inc., Bloomington IL, USA)
Procedure: Endorectal Advancement Flap — Surgical procedure for the treatment of anal fistula by an Advancement Mucosa Flap
  Other Names: Advancement Mucosa Flap

SUMMARY:
The purpose of this study is to determine whether anal fistula plug or endorectal advancement flap is more successful in the treatment of anal fistulas and compared both procedures with regards to cost.

DETAILED DESCRIPTION:
A detailed analysis will be performed to determine independent predicting factors of recurrence and of higher costs.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or more)
* Single anal fistula
* Surgically treated with anal fistula plug or endorectal advancement flap

Exclusion Criteria:

* Children or adolescents
* Pregnancy
* Patients treated with setons alone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2007-05; Primary Completion 2013-09 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Anal fistula recurrence rate | One year

SECONDARY OUTCOMES:
Cost | 3 days
  In-hospital costs. Typically 1 to 3 days of hospitalization
Complication rate | 3 days
  Classified according to the Clavien-Dindo Classification of Surgical Complications.
Length of hospital stay | 3 days
  Typically 1 to 3 days of hospitalization.
Independent factors predicting fistula recurrence | One year
  Multivariate analysis of parameters derived from patient demographics and characteristics, surgical procedure, and perioperative management.
Independent factors predicting higher costs | One year
  Multivariate analysis of parameters derived from patient demographics and characteristics, surgical procedure, and perioperative management.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver M Fisher, MD, Principal Investigator — University of Zurich; Antonio Nocito, MD, Study Chair — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Adamina M, Hoch JS, Burnstein MJ. To plug or not to plug: a cost-effectiveness analysis for complex anal fistula. Surgery. 2010 Jan;147(1):72-8. doi: 10.1016/j.surg.2009.05.018. Epub 2009 Sep 6. PMID 19733880
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912